CLINICAL TRIAL: NCT03978377
Title: Cardiopulmonary Toxicity of Thoracic Radiotherapy
Acronym: CLARIFY
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: CLARIFY
Record Dates: First submitted 2019-02-01; First posted 2019-06-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Oesophageal Cancer; Non Small Cell Lung Cancer
Keywords: Radiotherapy; Pulmonary hypertension
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Radiotherapy improves locoregional control and survival of thoracic tumour patients. However, the associated exposure of normal tissues, often leads to side effects and possibly even reduces survival. Indeed, there is growing evidence that overall survival after radiotherapy for lung and oesophageal cancer is related to the radiation dose to heart and lungs. This suggests that thoracic radiotherapy causes mortality, which is currently not recognized as radiation-induced toxicity. So the question arises how to explain this treatment-related mortality.

Interestingly, Ghobadi et al demonstrated in rats that thoracic irradiation can lead to pulmonary hypertension (PH). Histopathological analysis showed that radiation-induced PH closely resembles the pulmonary arterial hypertension (PAH) subtype. Moreover, in a clinical pilot study we confirmed early signs of PH including dose-dependent reductions in blood flow towards the lungs in radiotherapy patients.

In general PH significantly affects survival. Moreover, the PAH subtype is the most-rapidly progressive and lethal subtype. However, medical treatment can significantly slow down PAH progression, providing opportunities for secondary prevention. Yet, hard evidence that radiation-induced PH is a clinically relevant phenomenon in patients treated for thoracic tumours, is lacking.

DETAILED DESCRIPTION:
In the present study, the incidence and time course of treatment-related changes in cardio-pulmonary physiology will be assessed using standard diagnostic tools such as echocardiography, cardiac MRI (CMR) and serum biomarkers and relate them to the radiation dose distribution. Such insight in the characteristics of this possible radiation-induced PH and contributing risk factors is essential to develop primary (radiation dose optimization) prevention strategies.

The general objective of this study is to test the hypothesis that pulmonary hypertension (PH) is a clinically relevant radiation-induced side effect of thoracic irradiation. If confirmed this allows us to take appropriate measures in patient care to improve quality of life in thoracic cancer patients.

To investigate this hypothesis, the following specific aims have been defined:

* To assess the incidence and time course of PH in a prospective cohort study in patients treated with radiotherapy for lung or oesophageal cancer.
* To characterize other changes in myocardial function and pulmonary arteries, and their function using cardiac MR.
* To determine treatment-related risk factors, in particular radiation dose factors to the lungs and heart that could be used for future optimization strategies to minimize the risk of inducing PH in these patients.
* To determine the clinical impact by correlating PH to patient-rated outcome measure (PROMs) and survival. Taken together this study will determine if radiation-induced pulmonary hypertension is a clinically relevant toxicity and will provide information required for future studies on its prevention and treatment. In addition, more insight will be obtained on other forms of cardiovascular damage and complications that may occur in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oesophageal cancer in the mid or distal oesophagus and patients with NSCLC stage IIA-III or NSCLC stage IV with limited brain metastases (treatable with surgery or stereotactic radiosurgery) or SCLC limited disease (stage I-IIIB)
* Scheduled for external-beam radiotherapy with curative intention.
* WHO 0-2.
* Age >= 18 years
* Written informed consent.

Exclusion Criteria:

* No heart failure in the last 2 months
* No pulmonary embolism in the last 2 months
* COPD gold IV
* BMI >35
* History of thoracic radiotherapy
* Noncompliance with any of the inclusion criteria - For MRI part: Contra indications for MRI

For MRI part:

• contra-indications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study focuses on two patient populations: 1) Patients with oesophageal cancer in the mid or distal oesophagus, who will be treated with radiotherapy with curative intent, with or without chemotherapy, with or without surgery.
  2) Patients with NSCLC stage IIA-III or NSCLC stage IV with limited brain metastases (treatable with surgery or stereotactic radiosurgery) or SCLC limited disease (stage I-IIIB), who will be treated with radiotherapy with curative intent, with or without chemotherapy.
  Patients will be included in 3 participating centers:
  * University Medical Center Groningen, Groningen, The Netherlands
  * Beatson West of Scotland Cancer Centre /NHS Greater Glasgow and Clyde, Glasgow, United Kingdom
  * Radboud UMC, Nijmegen, The Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with high risk of pulmonary hypertension | 1 year
  High-risk pulmonary hypertension according to ESC/ERS classification

SECONDARY OUTCOMES:
Troponine T change | 1 year
  Change in Troponine T concentration, between baseline and at 1 year
NTproBNP change | 1 year
  Change in NTproBNP concentration, between baseline and at 1 year
Number of patients with intermediate risk of pulmonary hypertension | 1 year
  Intermediate risk of pulmonary hypertension according to ESC/ERS classification
Cumulative incidence of other late cardiopulmonary toxicity, as classified by CTCAE4.0 | 1 year
  Cumulative incidence of other late cardiopulmonary toxicity, as classified by CTCAE4.0
EORTC quality of life questionnaire C30 | 1 year
  PROMs (EORTC QoL C30), including five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting),
EORTC quality of life questionnaire LC13 | 1 year
  PROMs (EORTC QoL LC13), including lung cancer-associated symptoms (cough, haemoptysis, dyspnoea and site specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy and alopecia) and pain medication.

CONTACTS AND LOCATIONS:
Locations (3):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Radboud UMC, Nijmegen, Gelderland, Netherlands
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No